CLINICAL TRIAL: NCT05975723
Title: Effect of MIND Diet Intervention on Cognitive Function in Adults With Mild Cognitive Impairment
Brief Title: MIND Diet and Cognitive Function in Adults With MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Changzheng Yuan, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AARG-22-928604
Record Dates: First submitted 2023-07-13; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Mild Cognitive Impairment; Cognitive Function; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIND diet intervention (Experimental): Participants in the MIND diet group will receive an education program on a localized MIND diet for 1-year, and will be routinely followed up and given advice on other healthy lifestyles.
  Interventions: Behavioral: MIND diet education; Behavioral: Routine follow-up and general advice
- Control group (Active Comparator): Participants in the control group will be routinely followed up and given general advice on healthy lifestyle.
  Interventions: Behavioral: Routine follow-up and general advice

INTERVENTIONS:
Behavioral: MIND diet education — An intensified education program following a localized modified MIND diet for 1 year, which recommends 11 brain healthy food groups (green leafy vegetables, dark red and yellow vegetables, other vegetables, nuts, berries, beans, whole grains, seafood, poultry, olive/tea-seed oil and green tea) and limits intake of 4 unhealthy food groups (red meat and products, animal oil, pastries and sweets, and fried/fast food).
  Arms: MIND diet intervention
Behavioral: Routine follow-up and general advice — Routine follow-up administered by trained staff.

SUMMARY:
To examine the effects of a 1-year cluster-randomized controlled intervention of MIND diet on cognitive function among 240 participants with mild cognitive function (MCI) aged 50 years and above from 4 communities.

DETAILED DESCRIPTION:
The current study is a 1-year cluster-randomized controlled intervention trial designed to examine whether the a localized modified Mediterranean-Dietary Approaches to Stop Hypertension (DASH) dietary intervention for neurodegenerative delay (MIND) diet will improve cognitive function among 240 participants with MCI from 4 communities. The modified MIND diet recommends 11 brain healthy food groups (green leafy vegetables, dark red and yellow vegetables, other vegetables, nuts, berries, beans, whole grains, seafood, poultry, olive/tea-seed oil and green tea) and limits intake of 4 unhealthy food groups (red meat and products, animal oil, pastries and sweets, and fried/fast food). This study will randomly assign 240 MCI participants to two groups: A) MIND diet intervention group and B) control group, and estimate the cognitive and biological impacts of the 1-year intervention.

ELIGIBILITY:
Inclusion Criteria:

* At risk of cognitive decline: cognitive performance at the mean level or slightly lower than expected for age with no dementia (AD8>=3 and/or 5-min MoCA < 11)
* Free of physical disabilities that preclude participation in the study
* Willing to complete all study-related activities for 24 months
* Willing to be randomized to either intervention group

Exclusion Criteria:

* Allergic to more than one type of food (nuts, berries, olive oil, or fish)
* Diagnosed of dementia, severe diabetes mellitus, cardiovascular disease, cancer, thyroid disease, kidney disease, or liver disease
* Diagnosed of major depression or other neuropsychological diseases
* Severe loss of vision, hearing or communicative ability
* Substance abuse within 6 months or heavy alcohol consumption (> 2 drinks/day for women; > 3 drinks/day for men).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Global Cognition measured by comprehensive Neuropsychological Test Battery (NTB) | Up to one year
  Global cognitive performance (composite z-score) measured by comprehensive Neuropsychological Test Battery (NTB). The z-score calculation will use the population mean and standard deviation, and a higher z-score indicates better cognitive performance.
Change in Domain-specific Cognition | Up to one year
  NTB domain-specific cognitive performance (composite z-score) for memory, executive function, attention, language, visuomotor speed and visuoconstruction. The z-score calculation will use the population mean and standard deviation, and a higher z-score indicates better cognitive performance.

SECONDARY OUTCOMES:
Change in Clinical Dementia Rating-Sum of Boxes (CDR-SB) | Up to one year
  The Clinical Dementia Rating-Sum of Boxes (CDR-SB) is scored from 0 to 18. Higher scores reflect worse performance.
Change in Alzheimer's Disease Cooperative Study Activities of Daily Living Mild Cognitive Impairment-Activities of Daily Living Inventory (ADCS MCI-ADL) | Up to one year
  The Alzheimer's Disease Cooperative Study Activities of Daily Living-Mild Cognitive Impairment-Activities of Daily Living Inventory (ADCS MCI-ADL) is scored from 0 to 53. Higher scores reflect better performance.
Change in Pittsburgh Sleep Quality Index (PSQI) | Up to one year
  The Pittsburgh Sleep Quality Index (PSQI) is scored from 0 to 21. Higher scores indicate worse sleep quality.
Change in Montreal Cognitive Assessment (MoCA) score | Up to one year
  MoCA will be assessed to determine cognitive change.

OTHER OUTCOMES:
Change in dietary behaviour measured using a food frequency questionnaire | Up to one year
  To evaluate the behavioural effect of dietary changes of the MIND diet intervention package.
  Exploratory aim 1b: Changes in plasma levels of carotenoids, fatty acids, and vitamins (including folic acid). To evaluate the effect on nutritional biomarkers of the MIND diet intervention.
Change in depressive status measured using the Geriatric Depression Scale (GDS) | Up to one year
  To evaluate the effect on the depressive status of the MIND diet intervention. A higher GDS score indicates more severe depressive symptoms.
Change in anxiety status measured using the General Anxiety Disorder-7 (GAD-7) | Up to one year
  To evaluate the effect on the anxiety status of the MIND diet intervention. A higher GAD-7 score indicates more severe anxious symptoms.
Changes in plasma metabolic profiles measured using metabolome analysis | Up to one year
  To evaluate the effect on plasma metabolites of the MIND diet intervention. We will assay the metabolome using liquid chromatography-mass spectrometry (LC-MS) and construct an overall metabolic score of the diet as the outcome.
Changes in plasma inflammatory biomarkers | Up to one year
  To evaluate the effect on systematic inflammation of the MIND diet intervention. We will assay interferon-γ, Interleukin (IL)-10, IL-12p70, IL-13, IL-1β, IL-2, IL-4, IL-6, IL-8, Tumor Necrosis Factor alpha, and C-Reaction Protein and construct an overall plasma inflammatory biomarker score as the outcome.
Changes in the intestinal microbiome | Up to one year
  To evaluate the effect on intestinal microbiome biodiversity and abundance in specific species in faecal samples of the MIND diet intervention. We will assay microbiome using 16-S ribosomal RNA (rRNA) sequencing and construct an overall intestinal microbiome score as the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Changzheng Yuan, ScD, Study Chair — Zhejiang University
Locations (1):
- Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
When applicable, electronic data will be made available after trial completion.
Supporting Information: CSR
Time Frame: When the final research data published, the data and other related resources would be shared in the Global Alzheimer's Association Interactive Network (GAAIN).
Access Criteria: Review & Approval by the Publications and Presentation Committee.

REFERENCES:
- [Background] Chen H, Dhana K, Huang Y, Huang L, Tao Y, Liu X, Melo van Lent D, Zheng Y, Ascherio A, Willett W, Yuan C. Association of the Mediterranean Dietary Approaches to Stop Hypertension Intervention for Neurodegenerative Delay (MIND) Diet With the Risk of Dementia. JAMA Psychiatry. 2023 Jun 1;80(6):630-638. doi: 10.1001/jamapsychiatry.2023.0800. PMID 37133875
- [Background] Huang L, Tao Y, Chen H, Chen X, Shen J, Zhao C, Xu X, He M, Zhu D, Zhang R, Yang M, Zheng Y, Yuan C. Mediterranean-Dietary Approaches to Stop Hypertension Intervention for Neurodegenerative Delay (MIND) Diet and Cognitive Function and its Decline: A Prospective Study and Meta-analysis of Cohort Studies. Am J Clin Nutr. 2023 Jul;118(1):174-182. doi: 10.1016/j.ajcnut.2023.04.025. Epub 2023 Apr 25. PMID 37105521
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Liu X, Morris MC, Dhana K, Ventrelle J, Johnson K, Bishop L, Hollings CS, Boulin A, Laranjo N, Stubbs BJ, Reilly X, Carey VJ, Wang Y, Furtado JD, Marcovina SM, Tangney C, Aggarwal NT, Arfanakis K, Sacks FM, Barnes LL. Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) study: Rationale, design and baseline characteristics of a randomized control trial of the MIND diet on cognitive decline. Contemp Clin Trials. 2021 Mar;102:106270. doi: 10.1016/j.cct.2021.106270. Epub 2021 Jan 9. PMID 33434704